CLINICAL TRIAL: NCT00719121
Title: Placebo-Controlled, Investigator Blinded, Explorative Trial to Evaluate the Anti-inflammatory Effect of Multiple Topical Applications of R115866 Gel (0.35%) in Two Models of Cutaneous Inflammation in Healthy Male Subjects
Brief Title: Study on Anti-inflammatory Effects of Topical R115866 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: BT0700-107-BEL
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2008-07

CONDITIONS: Cutaneous Inflammation
MeSH Terms: conditions — Dermatitis | interventions — R 115866; Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (No Intervention): No Treatment
- B (Active Comparator): R115866 (0.35% gel)
  Interventions: Drug: Talarozole
- C (Active Comparator): R115866 Vehicle gel
  Interventions: Drug: Talarozole
- D (Active Comparator): Differin™, 0.1% adapalene gel
  Interventions: Drug: Differin™, 0.1% adapalene gel

INTERVENTIONS:
Drug: Talarozole — Topical Application (20 mg)
  Other Names: Rambazole, R115866
  Arms: B; C
Drug: Differin™, 0.1% adapalene gel — Topical Application (20 mg)
  Other Names: adapalene gel
  Arms: D

SUMMARY:
The purpose of this exploratory trial is to assess the anti-inflammatory effect(s) of topical R115866 in a model of UVB-induced inflammation and in a model of cutaneous irritation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index should be between 18 and 28 kg/m2
* Subjects are healthy as determined by medical history, physical examination and clinical laboratory tests carried out at screening
* Subjects with a phototype III or IV (according to Fitzpatrick classification)

Exclusion Criteria:

* Subjects with history of or active alcohol or substance abuse problems.
* Known hypersensitivity to azoles, adapalene, retinoids or any other ingredient of the gels
* Subjects who have a laboratory value which, in the opinion of the investigator, is clinically-relevant out of the normal range
* Subjects with clinically relevant abnormal ECG-intervals or morphology of the ECG, QTc interval >450 ms
* Use of vitamin A (>1000 µg/day) or the use of concomitant medication, except paracetamol; All other medication must have been stopped at least 14 days before the first administration of gel)
* Subjects who have received an investigational product which is not a biological within the month preceding the screening visit; If the investigational product is a biological, a 3-month wash-out period is required.
* Use of ultraviolet light (including artificial UVA and UVB as well as excessive natural sun exposure) unless stopped at Visit 1
* Subjects judged by the investigator to have a high probability of lack of compliance with the provisions of the protocol
* Subjects having any medical condition which, in the opinion of the investigator at the site, is a contraindication to enrollment

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint was the mean value of TEWL (Trans-epidermal water loss) | Day 1 through Day 9 of treatment

SECONDARY OUTCOMES:
Erythema | Day 1 through Day 8 of treatment and Day 15 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. G. Piérard, MD, PhD, Principal Investigator — Department of Dermatopathology Centre Hospitalier Universitaire du Sart-Tilman
Locations (1):
- Department of DermatopathologyCentre Hospitalier Universitaire du Sart Tilman, Liège, Belgium